CLINICAL TRIAL: NCT02767531
Title: Orlistat for the Treatment of Type I Hyperlipoproteinemia
Acronym: T1HLP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Abhimanyu Garg, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 012013-042
Record Dates: First submitted 2016-05-02; First posted 2016-05-10 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hyperlipoproteinemia Type I; Hypertriglyceridemia
MeSH Terms: conditions — Hyperlipoproteinemia Type I; Hypertriglyceridemia | interventions — Orlistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orlistat (Experimental): 120 mg of Orlistat will be given 3 times to patients weighing greater than 50 kg and patients weighing less than 40 kg will be given 60 mg of Orlistat 3 times a day for 3 months.
  Interventions: Drug: Orlistat
- Off drug (No Intervention): Standard therapy will be given for three months

INTERVENTIONS:
Drug: Orlistat — Orlistat is a gastric and pancreatic lipase inhibitor that is approved by the FDA for weight loss. It is available over-the-counter as 60 mg tablets under the trade name Alli, and available by prescription as 120 mg capsules under the trade name Xenical.
  Other Names: Alli
  Arms: Orlistat

SUMMARY:
Patients with Type I Hyperlipoproteinemia (T1HLP) have a rare form of hypertriglyceridemia marked by significant chylomicronemia and recurrent episodes of acute pancreatitis. T1HLP is caused by a deficiency of lipoprotein lipase or one of its cofactors. Many patients are a challenge to treat, as the only effective therapy available is an extremely low fat diet. This diet is exceedingly difficult to follow, and despite adherence, many patients still have chylomicronemia and develop acute pancreatitis.

Specific Aim: To determine the efficacy of a gastric and pancreatic lipase inhibitor, Orlistat, in reducing serum triglyceride levels in patients with T1HLP.

DETAILED DESCRIPTION:
Type I hyperlipoproteinemia is a rare, autosomal recessive metabolic disorder characterized by extreme hypertriglyceridemia due to a deficiency in lipoprotein lipase or related proteins. Treatment of these patients is challenging as triglyceride-lowering medications are ineffective. A low fat diet is helpful, however, despite good dietary compliance, some patients continue to have severe hypertriglyceridemia and recurrent pancreatitis which can be life threatening. Therefore, Investigator wish to investigate whether inducing dietary fat malabsorption or inhibiting chylomicron formation will cause further lowering of serum triglycerides (TG) beyond the effect of limiting dietary fat intake.

Investigator will study the efficacy and safety of an inhibitor of intestinal lipase (Orlistat) for reducing serum triglyceride levels in patients with Type I hyperlipoproteinemia. Investigator plan to enroll 20 patients with Type I hyperlipoproteinemia in a randomized, double-blind, placebo-controlled, cross-over trial. During the last week of each study period, fasting blood samples will be drawn for three consecutive days for serum lipids and chemistry panel. The primary endpoint will be serum triglycerides; the secondary endpoint variables will be fasting and postprandial serum chylomicron-TG levels, postprandial serum TG levels during a meal tolerance test and retinyl palmitate levels during a meal tolerance test. Repeated measures analysis of variance will be used for statistical comparisons.

These results may help in designing novel therapeutic approaches for patients with Type 1 hyperlipoproteinemia.

ELIGIBILITY:
Inclusion Criteria:

1. Type I hyperlipoproteinemia
2. Fasting serum triglyceride levels of greater than 1000 mg/dL
3. Age > 8 years

Exclusion Criteria:

1. Secondary hypertriglyceridemias due to diabetes, renal disease, hypothyroidism, alcoholism and drug therapy such as estrogens and estrogen analogues, steroids, HIVprotease inhibitors, retinoic acid derivatives and interferons
2. Pregnant or lactating women
3. Significant liver disease (elevated transaminases > 2 times upper limit of normal) Alcohol abuse (> 7 drinks or 84 g per week for women and > 14 drinks or 168 g per week for men)
4. Severe anemia (hematocrit < 24%)
5. Drug use (cocaine, marijuana, LSD, etc.)
6. Major surgery in the past three months
7. Congestive heart failure
8. Serum creatinine greater than 2.5 mg/dL
9. Cancer within the past five years
10. Gastrointestinal surgery in the past
11. Current therapy with anti-coagulants, digoxin, and anti-arrhythmics
12. Current therapy with cyclosporine
13. Chronic malabsorption syndromes
14. Cholestasis
15. Acute illnesses such as acute pancreatitis in the last 8 weeks

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2015-12; Primary Completion 2018-05-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu Garg, MD, Principal Investigator — University of Texas
Locations (1):
- UT Southwestern Medical Center 5323 Harry Hines Blvd, Dallas, Texas, United States

REFERENCES:
- [Derived] Patni N, Quittner C, Garg A. Orlistat Therapy for Children With Type 1 Hyperlipoproteinemia: A Randomized Clinical Trial. J Clin Endocrinol Metab. 2018 Jun 1;103(6):2403-2407. doi: 10.1210/jc.2018-00369. PMID 29659879

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized,open-label, crossover trial with four periods and two sequences ("orlistat" and "off" for 3 months each) was conducted.
Groups:
- Orlistat Then Off Therapy: Randomized to Orlistat for first 3 months, then cross over to no therapy for 3 months, followed by repeat sequence of Orlistat for additional 3 months, and no therapy for next 3 months
- Off Orlistat Then Orlistat: Randomized to no therapy for first 3 months and then cross over to Orlistat for 3 months and then repeat sequence of no therapy for additional 3 months and then Orlistat for next 3 months
Period: Period 1
Arm/Group | Orlistat Then Off Therapy | Off Orlistat Then Orlistat
Started | 1 (Orlistat therapy) | 1 (Off Orlistat)
Completed | 1 | 1
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Orlistat Then Off Therapy | Off Orlistat Then Orlistat
Started | 1 (Off Orlistat) | 1 (Orlistat Therapy)
Completed | 1 | 1
Not Completed | 0 | 0
Period: Period 3
Arm/Group | Orlistat Then Off Therapy | Off Orlistat Then Orlistat
Started | 1 (Orlistat Therapy) | 1 (Off Orlistat)
Completed | 1 | 1
Not Completed | 0 | 0
Period: Period 4
Arm/Group | Orlistat Then Off Therapy | Off Orlistat Then Orlistat
Started | 1 (Off Orlistat) | 1 (Orlistat Therapy)
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Features of Patients Enrolled: 120 mg of Orlistat will be given 3 times to patients weighing greater than 50 kg and patients weighing less than 40 kg will be given 60 mg of Orlistat 3 times a day for 3 months.
  The patients were randomized to receive 3 months of orlistat or no therapy (off), then crossed over to the other arm, and this sequence was then repeated for an additional 6 months
Arm/Group | Baseline Features of Patients Enrolled
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
Triglyceride [Mean (Full Range); unit: mg/dL] | 1674 [1611 to 1737]

OUTCOME MEASURES:

1. Primary Outcome: Fasting Serum Triglycerides
Description: Fasting blood samples were collected on three consequetive days at the end of each three month period. Mean values of the three days were calculated.
Time Frame: 3 days
Population: The patients were randomized to receive 3 months of orlistat or no therapy (off), then crossed over to the other arm, and this sequence was then repeated. Because only 2 patients participated, the results are provided per sequence and not per intervention.
Measure: Mean (Full Range); unit: mg/dL
Groups:
- Orlistat and Then Off Therapy: Randomized to Orlistat for first 3 months, then cross over to no therapy for 3 months, followed by repeat sequence of Orlistat for additional 3 months, and no therapy for next 3 months
  120 mg of Orlistat will be given 3 times to patients weighing greater than 50 kg and patients weighing less than 40 kg will be given 60 mg of Orlistat 3 times a day for 3 months.
- Off Therapy and Then Orlistat: Randomized to no therapy for first 3 months and then cross over to Orlistat for 3 months and then repeat sequence of no therapy for additional 3 months and then Orlistat for next 3 months
Arm/Group | Orlistat and Then Off Therapy | Off Therapy and Then Orlistat
Number analyzed (Participants) | 1 | 1
mg/dL
  Period 1 | 705 [656 to 730] | 1827 [1266 to 2320]
  Period 2 | 1511 [1226 to 1750] | 1007 [964 to 1040]
  Period 3 | 758 [617 to 876] | 3121 [2780 to 3490]
  Period 4 | 1614 [1540 to 1680] | 1181 [1122 to 1248]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Orlistat: Each of the two patients, were randomized to receive Orlistat for 3 months in two periods.
  Patient 1 took Orlistat 60 mg with the first and second meal and 120 mg with the third meal, whereas Patient 2 took 60 mg of Orlistat 3 times daily with meals.
- Off Therapy: Each of the two patients, were randomized to "Off therapy" for 3 months in two periods.
Arm/Group | Orlistat | Off Therapy
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 0/2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orlistat (N=2) | Off Therapy (N=2)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0) — Patient1 had a mild increase in passage of gas and bloating, and patient 2 had constipation with mild stool leakage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT02767531/Prot_SAP_000.pdf